CLINICAL TRIAL: NCT04667312
Title: CODAK: A Retrospective Observational Research Study to Describe the Characteristics and Real-world Clinical Outcomes of Patients With Locally Advanced, Unresectable Stage III Non-small Cell Lung Cancer Receiving Durvalumab in the UK.
Brief Title: Observational Study of Durvalumab in Patients With Non-small-cell Lung Cancer in the United Kingdom
Acronym: CODAK
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4191R00038
Record Dates: First submitted 2020-11-27; First posted 2020-12-14 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Non-Small Cell Lung Cancer NSCLC
Keywords: NSCLC unresectable stage III
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Durvalumab — Durvalumab
  Other Names: Imfinzi

SUMMARY:
This is a retrospective observational research study to describe the characteristics and real-world clinical outcomes of patients with locally advanced, unresectable Stage III non-small cell lung cancer receiving durvalumab in the United Kingdom (the CODAK study). Physicians who have treated patients who have locally advanced, unresectable Stage III NSCLC with durvalumab will be requested to recruit patients to have their clinical data abstracted from their clinical records in line with local laws. Data from this study will provide UK-specific real-world data on patients receiving durvalumab through the Early Access Programme (EAP) or post-reimbursement.

DETAILED DESCRIPTION:
Primary Objectives

The primary study objectives, in patients with locally advanced, unresectable Stage III NSCLC treated with durvalumab as part of the UK EAP or non-EAP, are:

1. To describe clinical outcomes
2. To describe the patient demographic and clinical characteristics Secondary Objective

1. To describe treatment patterns of durvalumab

ELIGIBILITY:
Inclusion Criteria:

* Patient has documented diagnosis of locally advanced, unresectable Stage III NSCLC
* Patient has received platinum-based CRT and received ≥1 dose of durvalumab
* Patient was initiated on durvalumab (index event) between 1st September 2017 and 31st December 2019 via the EAP or non-EAP
* Patient was aged ≥18 years at durvalumab initiation

Exclusion Criteria:

* Patients who participated in the PACIFIC-R study
* Participation in any clinical study with an investigational product at the time of durvalumab initiation or during the observational period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is adult patients with locally advanced, unresectable Stage III NSCLC treated with durvalumab following platinum based chemoradiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 12 months
  This study will estimate the proportion of patients known to be alive at 12 months post-index event
Overall Survival | 24 months
  This study will estimate the proportion of patients known to be alive at 24 months post-index event

SECONDARY OUTCOMES:
Progression Free Survival | 12 months
  In this study, rwPFS will describe the proportion of patients known to be alive and free from disease progression at 12 months post-index event,
Progression Free Survival | 24 months
  In this study, rwPFS will describe the proportion of patients known to be alive and free from disease progression at 24 months post-index event,
Second Progression Free Survival | 12 months
  In this analysis, rwPFS2 describes the proportion of patients who progressed on durvalumab and who were known to be alive and had not progressed (including metastatic disease) on subsequent treatment at 12 months post-durvalumab initiation.
Second Progression Free Survival | 24 months
  In this analysis, rwPFS2 describes the proportion of patients who progressed on durvalumab and who were known to be alive and had not progressed (including metastatic disease) on subsequent treatment at 24 months post-durvalumab initiation.
Best Overall Response | Up to 24 months
  Best overall response, as recorded in medical records, will be described as complete response [CR], partial response [PR], stable disease [STD], absence of progression, progressive disease [PD], death, not recorded [NR]).
Time to Treatment Discontinuation | Up to 24 months
  Time from date of durvalumab initiation to date of discontinuation will be summarized using the Kaplan-Meier method, including the presentation of Kaplan-Meier plots.
Time to first subsequent therapy | Up to 24 months
  Time to initiation of first subsequent therapy will be summarized using the Kaplan-Meier method, including the presentation of Kaplan-Meier plots.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Franks, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (10):
- United Kingdom (10):
  - East Kent Hospital, Canterbury
  - Velindre Hospital, Cardiff
  - Harrogate and district NHS foundation Trust, Harrogate
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Guy's Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation, Manchester
  - Queen Alexandra Hospital, Portsmouth
  - Musgrove Park Hospital, Taunton
  - Royal Cornwall Hospitals NHS Trust, Truro

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis 20Sep2023 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4191R00038&attachmentIdentifier=8667ed8a-a98b-45a2-864c-577d46155d72&fileName=D4191R00038_CODAK_Study_Synopsis_Trial.Gov_20Sep23_.pdf&versionIdentifier=